CLINICAL TRIAL: NCT06240416
Title: A Randomized Clinical Trial Comparing Autogenous Particles Harvesting During Implant Surgery Using Low-speed Drilling Without Irrigation and High-speed Drilling With Irrigation
Brief Title: Autogenous Particles Harvesting During Implant Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26302019
Record Dates: First submitted 2024-01-09; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-12

CONDITIONS: Dental Implant Failed
Keywords: Dental implants; Osteotomy; Temperature; Histology
MeSH Terms: interventions — Therapeutic Irrigation

STUDY DESIGN:
Intervention Model Description: A split mouth randomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): High speed drilling (800 rpm) with irrigation
  Interventions: Procedure: High speed drilling with irrigation
- Test group (Experimental): Low speed drilling (50 rpm) without irrigation
  Interventions: Procedure: Low speed drilling without irrigation

INTERVENTIONS:
Procedure: Low speed drilling without irrigation — Low-speed drilling (50 rpm) irrigation to perform the osteotomy
  Arms: Test group
Procedure: High speed drilling with irrigation — High-speed drilling (800 rpm) irrigation to perform the osteotomy
  Arms: Control group

SUMMARY:
The aim was to compare the osteoblast activity and osteogenic potential of autogenous bone particles harvested using three different techniques, determine the most advantageous method of collecting autogenous bone particles.

Bone particles were harvested during dental implant surgery using low-speed drilling and high speed drilling. After the osteoblasts were cultured, cell proliferation, migration, mineralization, transcription of osteogenesis-related genes, secretion of osteogenesis-related proteins, and osteoinductive protein content in the bone particle matrix were evaluated

DETAILED DESCRIPTION:
A total of 60 individual dental implants will be placed in this study. Each patient will receive two dental implants (Spain), each measuring 10 mm in length and 4 mm in diameter, for the replacement of missing teeth in the right and left mandibular first molars. The surgery will be performed under local anesthesia (0.5% articaine with epinephrine) with the elevation of a mucoperiosteal flap. For the randomization of the implant osteotomy milling protocol in each hemimandible, an online randomization service (www.randomization.com) will be utilized.

In each patient, the conventional high-speed milling protocol with irrigation using physiological saline will be employed in one hemimandible. In the other hemimandible, the implant osteotomy will be performed using a low-speed milling protocol without irrigation.

The milling sequence for the conventional high-speed milling protocol with irrigation will be as follows: the osteotomy will be initiated with a 2.0 mm diameter marking drill, followed by a pilot drill of the same diameter. Subsequently, drills of 2.6/3.2/ and 3.6 mm diameters will be used consecutively. All drills will be used at a speed of 800 rpm and at a depth of 10 mm.

On the other hand, the milling sequence for the low-speed milling protocol without irrigation will be the same, but all drills will be used at a speed of 50 rpm (at the same depth of 10 mm). Finally, once the dental implant and closing screw are inserted, the mucoperiosteal flap will be sutured with simple stitches using synthetic polyamide suture, without immediate prosthetic loading. In all cases, postoperative medication will include 500 mg/8 h amoxicillin for 7 days (in cases of penicillin allergy, 300 mg/8 h clindamycin for 7 days), and 600 mg/8 h ibuprofen for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Legal age
* Informed consent signed
* Bilateral mandibular dental absence of 3.6 and 4.6 for more than 3 months
* Normal bone density in the posterior mandibular sector with type II/III bone (range of 500-850 HU) according to the classification of Norton and Gamble
* No medical contraindications for the performance of oral surgical procedures (ASA I/II).

Exclusion Criteria:

* Presence of any disease, condition, or medication that may compromise the healing and/or osseointegration of dental implants (such as diabetes mellitus, bisphosphonate administration, or severe osteoporosis)
* Presence of any severe mental disorder
* Patients who have undergone head and neck radiotherapy in the previous 18 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2024-04-05 (Estimated); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Study of the size of bone particles collected during implant osteotomy, the presence or absence of collagen fibrils, and the levels of calcium and phosphorus in them. | day 1
  Once the amount of collected bone has been analyzed, 100 mg of bone will be used for the remaining study variables.
  The bone samples will be embedded in a 37% phosphoric acid gel for 15 seconds and then washed with plenty of water to remove the remaining acid. Subsequently, the samples will be mounted on holders for examination under the scanning electron microscope after receiving a carbon coating.
  After visualizing the samples at 100X, digital images will be taken for analysis using the image analysis software ImageJ.
  Finally, calcium and phosphorus levels will be analyzed using the Inca Microanalysis Systems software.
  The size will be expressed in nm.

SECONDARY OUTCOMES:
Quantify BMP-2 and VEGF in the bone collected during implant osteotomy using conventional and low-speed milling. | day 14
  The sterile Eppendorf tubes containing 100 mg of collected bone with one of the two compared protocols will be centrifuged at 217 g for 6 minutes. The supernatant will be collected and used to quantify BMP-2 and VEGF using an ELISA kit. The procedure will be carried out following the protocol provided by the manufacturer. Absorbance at 405 nm will be measured using an EXL-800 type ELISA reader.
  The variable will be expressed in % per 100mg
Analysis of the morphology and number of osteoblasts in the bone collected during implant osteotomy. | day 14
  To compare the morphology and number of osteoblasts in the bone collected during the milling sequence with the two compared protocols, the 100 mg of bone will be immediately cultured in α-MEM supplemented with fetal bovine serum and 1% antibiotic (penicillin 10,000 U/ml and streptomycin 10,000 µg/ml) The culture medium will be changed every 3 days.
  The morphology and number of cultured osteoblasts will be observed at 7 and 14 days. After visualization under a 40X optical microscope, the morphology will be described as normal or abnormal.
  The variable will be expressed in % per 100mg
Assessment of the presence of precipitated calcium nodules in the cell culture of osteoblasts after collecting bone during implant osteotomy. | day 21
  To compare the possible presence of precipitated calcium nodules in the cell culture of osteoblasts after collecting bone during the milling sequence with the two compared protocols, we will use the fourth passage of cultured osteoblasts (at 21 days of cultivation). Cells will be washed with PBS, fixed with 75% cold ethanol for 1 hour, and incubated with 1 ml of 0.1% alizarin red at pH 8.3 (Sigma-Aldrich Quimica S.A., Madrid, Spain) for 10 minutes. Then, if there are precipitated calcium nodules, they will be stained red and observed under the optical microscope. Finally, we will use a solution of 20% methanol and 10% acetic acid for 10 minutes to dissolve the alizarin red. Results will be expressed qualitatively by measuring absorbance at 550 nm using an EXL-800 type ELISA reader.
  The variable will be expressed in %
Study of cell viability (cell proliferation assay) | day 12
  We will also use the fourth passage of cultured osteoblasts (at 21 days of cultivation). The cells will be seeded in 96-well culture plates at a density of 1 X 103 cells per well. Cell proliferation will be assessed at 2, 6, and 12 days of incubation using the 3-(4,5-dimethylthiazol-2-yl)-2,5-diphenyl-2H-tetrazolium bromide (MTT) assay. First, 20 µl of MTT (Sigma-Aldrich Quimica S.A., Madrid, Spain) will be added to the medium and incubated for 4 hours. Subsequently, we will remove the medium and add 150 µl of dimethyl sulfoxide (Sigma-Aldrich Quimica S.A., Madrid, Spain) to each well. The results will be analyzed by measuring absorbance at 490 nm.
  The variable will be expressed in %
Determination of the cell cycle (G0/G1, G2/M, and S) | day 21
  For the study of the cell cycle, we will also use the fourth passage of cultured osteoblasts (at 21 days of cultivation). Cells will be detached from the cell culture flasks using 0.05% trypsin (Sigma-Aldrich Quimica S.A., Madrid, Spain) and 0.02% EDTA. Afterward, they will be washed and suspended in PBS for cell cycle analysis. The cells will be incubated at 37º C for 30 minutes with 100 ml of RNase (1 mg/ml) and 100 ml of propidium iodide.
  The DNA content of the stained cells will be studied using a FACSCaliburTM flow cytometer with a 488 nm argon laser to collect forward scatter (FSC), side scatter (SSC), and propidium iodide fluorescence intensity (PLA-2) data from 2000 events. The data will be analyzed using the CELLQUEST software and the MODFIT program, determining the percentage of cells in G0/G1, G2/M, and S phases.
  The variable will be expressed in %
Assessment of cell migration capability | day 1
  For the study of cell migration capability, we will also use the fourth passage of cultured osteoblasts (at 21 days of cultivation). Cells will be seeded in 6-well culture plates at a density of 5 X 104 cells per well and incubated for 24 hours to reach 100% confluence. Subsequently, 3 parallel lines will be drawn in each well using a sterile 300 µl pipette tip to create empty cell spaces, and cell migration will be observed at 6, 12, and 24 hours.
  Cell migration will be determined using the MIP-4.5 image analysis system. Using digital images of each well at 6, 12, and 24 hours, 10 lines of separation/approach of the empty cell spaces will be measured, and the distance traveled by the cells will be calculated using the formula: migration distance = (A0/2) - (At/2), where A0 is the initial width of the cell-free space, and At is the width of the cell-free space at 6, 12, or 24 hours.
  The variable will be expressed in %
Analysis cell viability ratios in the bone collected during implant osteotomy. | day 14
  Cell viability ratios of osteoblasts will be studied on day 14. Cells will be separated from the cell culture flasks using 0.05% trypsin (Sigma-Aldrich Quimica S.A., Madrid, Spain) and quantified using a Neubauer chamber. Then, cells will be stained with trypan blue to determine cell viability ratios.
  The variable will be expressed in % per 100mg

IPD SHARING:
Plan to Share IPD: Undecided